CLINICAL TRIAL: NCT04957134
Title: The Efficacy and Safety of Electro-acupuncture for Abdominal Obesity: Original Study for a Multicenter, Randomized, Sham-controlled Trial
Brief Title: Efficacy of Electro-acupuncture for Abdominal Obesity: Study for a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wang Jian, Hubei Provincial Hospital of Traditional Chinese Medicine, Hubei Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZY2021Z004
Record Dates: First submitted 2021-06-24; First posted 2021-07-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Abdominal
Keywords: Abdominal obesity; Electro-acupuncture; Randomized controlled trial
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture (Experimental): Participants will receive electro-acupuncture combined with lifestyle intervention. Participants will receive the treatment of electroacupuncture 3 times a week to fulfill a 8-session treatment course.
  Interventions: Device: Electro-acupuncture
- Sham electro-acupuncture (Placebo Comparator): Participants will receive the treatment of sham electro-acupuncture 3 times a week to fulfill a 8-session treatment course, A superficial skin penetration (2-3 mm in depth) at nonacupoints will be performed in the sham acupuncture group, without needle manipulation for De qi. The internal output power cord of the electrical acupuncture stimulation instrument is interrupted.
  Interventions: Device: Sham electro-acupuncture

INTERVENTIONS:
Device: Electro-acupuncture — The acupoints of electro-acupuncture will be selected as Zusanli ,Sanyinjiao ,Zhongwan , Tianshu , Shuifen , Daheng ,Daimai , Shuidao ,Huaroumen and Fujie . We will deliver electrical stimulation with dense-disperse waves at 50 Hz and 10 V through the electrical acupuncture stimulation instrument to the abdominal points. The bodily needles will be retained for 30 minutes . Electro-acupuncture treatment will be applied 3 times a week, once every other day, for 8 consecutive weeks.
  Arms: Electro-acupuncture
Device: Sham electro-acupuncture — The acupoints of sham electro-acupuncture will be selected as nonacupoints . The internal output power cord of the electrical acupuncture stimulation instrument will be interrupted. The bodily needles will be retained for 30 minutes . Sham acupuncture treatment will be applied 3 times a week, once every other day, for 8 consecutive weeks.
  Arms: Sham electro-acupuncture

SUMMARY:
Electro-acupuncture provides stimulation to acupoints, and has been widely used to treat abdominal obesity in China despite of lack of high-level evidence for treatment efficacy. The study will investigate whether the electroacupuncture can alleviate clinical symptoms and the mechanism of action in patients with abdominal obesity.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial from May 2021 to December 2022, including 68 participants with abdominal obesity. The participants will be randomly divided into 2 groups in a 1:1 allocation ratio.The intervention group will receive electroacupuncture; the control group will receive sham acupuncture. Each treatment will last 12 weeks, including 8 weeks of intervention period and 24 weeks of follow-up. The primary outcome is the waist circumference (WC), the secondary outcomes include weight, body mass index (BMI), hipline, waist-hip-ratio (WHR), Insulin resistance index (IRI), blood fat, metabolomics will be used analysis the mechanism. The adverse events will be recorded during the intervention and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited for this study should meet the following inclusion criteria:

  1.Satisfying the criteria for the diagnosis of abdominal obesity; 2.18 years old≤age≤55 years old; 3.Being able to fully understand and voluntarily sign informed consent.

Exclusion Criteria:

* Patients with any of the following criteria will be excluded from the study:

  1. Presence of endocrine disorders such as: polycystic ovary syndrome; Cushing's syndrome; uncorrected thyroid disease.
  2. Presence of diabetes mellitus, or hypertension, or abnormal liver and kidney functions, or mental diseases.
  3. Pregnant or lactating state, women who plan to become pregnant within 12 weeks.
  4. History of bulimia, anorexia, or any other eating disorders.
  5. Use of medications in the past 3 months, such as diet drugs, corticosteroids, antidepressants, which may affect weight or appetite.
  6. History of surgical weight loss, postoperative adhesions.
  7. History of participating in a clinical study of weight loss or any other therapies to lose weight in the past 3 months.
  8. Unable to cooperate with the research caused by other diseases or reasons.
  9. Received acupuncture within 6 months before enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline waistline at 8 weeks. | week 0,week 4,week 8,week 20,week 32
  Waistline will be measured around the abdomen at the level of the umbilicus (belly button).

SECONDARY OUTCOMES:
Change from baseline body weight at 8 weeks. | week 0,week 4,week 8,week 20,week 32
  Body weight will be measured by a body composition analyzer (OMRON V.BODY).
Change from baseline body mass index at 8 weeks. | week 0,week 4,week 8,week 20,week 32
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Change from baseline the body fat percentage at 8 weeks. | week 0,week 8,week 32
  The body fat percentage (BFP) of a human or other living being is the total mass of fat divided by total body mass, multiplied by 100. Body fat percentage will be measured by a body composition analyzer (OMRON V.BODY).
Change from baseline hip circumference at 8 weeks. | week 0,week 4,week 8,week 20,week 32
  Hip circumference will be measured at the level of maximum posterior extension of the buttocks.
Change from baseline waist-to-hip ratio at 8 weeks. | week 0,week 4,week 8,week 20,week 32
  Waist-to-hip ratio is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement ( W ÷ H ).
Changes from baseline insulin resistance index at 8 weeks. | week 0, week 8
  Examined with the blood sample.
Changes from baseline blood fat at 8 weeks. | week 0, week 8
  Examined with the blood sample.
Changes from baseline blood pressure at 8 weeks | week 0,week 4,week 8,week 32
  Both Systolic and diastolic blood pressure assessed by office and ambulatory blood pressure monitoring(mmHg).
Changes from baseline the IWQOL - Lite scale score at 8 weeks | week 0,week 8,week 32
  Quality of life was examined using the Impact of Weight on Quality of Life (IWQOL) questionnaire, which has a score range from 0(worst) to 100(best).
Changes from baseline the Kessler 10 scale at 8weeks. | week 0,week 8,week 32
  10 item self-report measure of psychological distress with five response categories (none of the time, a little of the time, some of the time, most of the time, all of the time). Scores range from 10 to 50; a higher score indicates more psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Zhou, Professor, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (1):
- Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The overall data outcome will be published in the form of public paper before december 2024.

REFERENCES:
- [Background] Carbone A, Al Salhi Y, Tasca A, Palleschi G, Fuschi A, De Nunzio C, Bozzini G, Mazzaferro S, Pastore AL. Obesity and kidney stone disease: a systematic review. Minerva Urol Nefrol. 2018 Aug;70(4):393-400. doi: 10.23736/S0393-2249.18.03113-2. Epub 2018 May 31. PMID 29856171
- [Background] Zhang N, Du SM, Ma GS. Current lifestyle factors that increase risk of T2DM in China. Eur J Clin Nutr. 2017 Jul;71(7):832-838. doi: 10.1038/ejcn.2017.41. Epub 2017 Apr 19. PMID 28422119
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Biemann R, Roomp K, Noor F, Krishnan S, Li Z, Shahzad K, Borucki K, Luley C, Schneider JG, Isermann B. Gene expression profile of CD14+ blood monocytes following lifestyle-induced weight loss in individuals with metabolic syndrome. Sci Rep. 2020 Oct 20;10(1):17855. doi: 10.1038/s41598-020-74973-2. PMID 33082492
- [Background] Lee JJ, Sundar KM. Evaluation and Management of Adults with Obstructive Sleep Apnea Syndrome. Lung. 2021 Apr;199(2):87-101. doi: 10.1007/s00408-021-00426-w. Epub 2021 Mar 13. PMID 33713177
- [Background] Viner RM, Hsia Y, Tomsic T, Wong IC. Efficacy and safety of anti-obesity drugs in children and adolescents: systematic review and meta-analysis. Obes Rev. 2010 Aug;11(8):593-602. doi: 10.1111/j.1467-789X.2009.00651.x. Epub 2009 Nov 17. PMID 19922432
- [Background] Chan EW, He Y, Chui CS, Wong AY, Lau WC, Wong IC. Efficacy and safety of lorcaserin in obese adults: a meta-analysis of 1-year randomized controlled trials (RCTs) and narrative review on short-term RCTs. Obes Rev. 2013 May;14(5):383-92. doi: 10.1111/obr.12015. Epub 2013 Jan 21. PMID 23331711
- [Background] Scheen AJ, Van Gaal LF. Combating the dual burden: therapeutic targeting of common pathways in obesity and type 2 diabetes. Lancet Diabetes Endocrinol. 2014 Nov;2(11):911-22. doi: 10.1016/S2213-8587(14)70004-X. Epub 2014 Feb 19. PMID 24731666
- [Background] Tronieri JS, Wadden TA, Walsh OA, Berkowitz RI, Alamuddin N, Gruber K, Leonard S, Chao AM. Effects of liraglutide plus phentermine in adults with obesity following 1 year of treatment by liraglutide alone: A randomized placebo-controlled pilot trial. Metabolism. 2019 Jul;96:83-91. doi: 10.1016/j.metabol.2019.03.005. Epub 2019 Mar 20. PMID 30902750
- [Background] Liang CM, Hu H, Wang CX, Sun SG, Yang WJ, Pan L. [Randomized Controlled Clinical Trials for Acupuncture Treatment of Abdominal Obesity]. Zhen Ci Yan Jiu. 2016 Apr;41(2):159-62, 174. Chinese. PMID 27323445
- [Background] Liang CM, Hu H, Li YY. [Acupuncture treatment of abdominal obesity patients by "belt vessel (Daimai) regulating method"]. Zhen Ci Yan Jiu. 2012 Dec;37(6):493-6. Chinese. PMID 23383460
- [Background] Zhang YJ, Li J, Huang W, Mo GY, Wang LH, Zhuo Y, Zhou ZY. [Effect of electroacupuncture combined with treadmill exercise on body weight and expression of PGC-1alpha， Irisin and AMPK in skeletal muscle of diet-induced obesity rats]. Zhen Ci Yan Jiu. 2019 Jul 25;44(7):476-80. doi: 10.13702/j.1000-0607.180460. Chinese. PMID 31368276
- [Background] Huang W, Chen X, Zhang Y, Wang L, Wang J, Zhang Y, Wei D, Zhou Z. Acupoint catgut embedding for obesity: A protocol of systematic review. Medicine (Baltimore). 2020 Dec 18;99(51):e23728. doi: 10.1097/MD.0000000000023728. PMID 33371124
- [Background] Chen X, Huang W, Wei D, Ding DG, Jiao Y, Pan HL, Jin YT, Zheng YW, Zhang YJ, Zhang YR, Liu YR, Zhou ZY. Clinical effect of catgut implantation at acupoints for the treatment of simple obesity: A multicentre randomized controlled trial. Medicine (Baltimore). 2020 Nov 25;99(48):e23390. doi: 10.1097/MD.0000000000023390. PMID 33235115
- [Background] Chen X, Huang W, Hu F, Jin YT, Hong ZH, Zhou ZY. [Regularity of Acupoint Selection for Simple Obesity Treated by Acupoint Catgut Embedding Based on Complex Network Technology]. Zhen Ci Yan Jiu. 2018 Sep 25;43(9):585-90. doi: 10.13702/j.1000-0607.170448. Chinese. PMID 30232869
- [Background] Gao Y, Wang Y, Zhou J, Hu Z, Shi Y. Effectiveness of Electroacupuncture for Simple Obesity: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2020 Jun 28;2020:2367610. doi: 10.1155/2020/2367610. eCollection 2020. PMID 32714399
- [Background] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Background] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Background] Zhang CY, Yang L. [Effect of Acupuncture Therapy on Visceral Fat Thickness in Simple Central Obesity Patients]. Zhen Ci Yan Jiu. 2015 Dec;40(6):484-8. Chinese. PMID 26887212
- [Background] Yu Z, Xia Y, Ju C, Shao Q, Mao Z, Gu Y, Xu B. Electroacupuncture regulates glucose-inhibited neurons in treatment of simple obesity. Neural Regen Res. 2013 Mar 25;8(9):809-16. doi: 10.3969/j.issn.1673-5374.2013.09.005. PMID 25206728
- [Background] Zhong LL, Kun W, Lam TF, Zhang SP, Yang JJ, Ziea TC, Ng B, Bian ZX. The combination effects of body acupuncture and auricular acupressure compared to sham acupuncture for body weight control: study protocol for a randomized controlled trial. Trials. 2016 Jul 25;17(1):346. doi: 10.1186/s13063-016-1458-2. PMID 27457720
- [Background] Matsueda K, Hongo M, Tack J, Saito Y, Kato H. A placebo-controlled trial of acotiamide for meal-related symptoms of functional dyspepsia. Gut. 2012 Jun;61(6):821-8. doi: 10.1136/gutjnl-2011-301454. Epub 2011 Dec 9. PMID 22157329
- [Derived] Chen X, Zhang Y, Fu C, Huang M, Wei D, Zhou W, Liu Y, Huang B, Rao Y, Zhang Y, Xia H, Hu Y, Li H, Huang W, Zhou Z. Electroacupuncture Reduces Waistline in Patients with Abdominal Obesity: A Randomized Controlled Trial with Mechanistic Analysis of Lipidomic and Intestinal Microbiota. Diabetes Metab Syndr Obes. 2025 Sep 30;18:3649-3669. doi: 10.2147/DMSO.S551806. eCollection 2025. PMID 41050180